CLINICAL TRIAL: NCT06266520
Title: Micro-needle-knife Therapy in Releasing the Superficial Fascia for Patients With Acute Ankle Sprain: an Assessor-blinded, Randomised Controlled Trial
Brief Title: MNK Therapy in Releasing the Superficial Fascia for Patients With AAS: an Assessor-blinded, Randomised Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sen-wei Lu (Other)
Responsible Party: Sponsor-Investigator, Sen-wei Lu, Prof., Affiliated Dongyang Hospital of Wenzhou Medical University
Organization: Affiliated Dongyang Hospital of Wenzhou Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DongyangH
Record Dates: First submitted 2024-02-06; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Acute Ankle Sprain
Keywords: acute ankle sprain; micro-needle-knife; superficial fascia; randomized controlled trial
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (MNK therapy to release the superficial fascia) (Experimental): The patient, positioned supine and wearing shorts for full lower limb exposure, undergoes layered palpation by the practitioner at the procedure points, identifying tender nodules and swelling in superficial fascia and muscles, followed by disinfection with an iodophor cotton swab. The practitioner, donning sterile latex gloves, holds the micro-needle-knife between the thumb and index finger of the right hand, inserting it parallel to the body's longitudinal axis, while the left thumb presses and holds the cord-like nodules for parallel incisions, with a maximum insertion depth of 5mm, performing lifting and cutting motions. Depending on the nodule size, 1-3 incisions are made. Post-procedure, any bruising or tissue fluid is expelled by massaging from distal to proximal around the incision. The area is then compressed with dry sterile gauze until bleeding ceases. Treatments are administered every other day, totaling six sessions.
  Interventions: Procedure: MNK therapy to release the superficial fascia
- Group 2 (acupuncture) (Active Comparator): Group 2 receives acupuncture treatment, employing needles produced by Suzhou Medical Supplies Factory Co., Ltd., with specifications of 0.30mm*40mm and conforming to standard GB2024-1994. Patients, positioned prone or laterally with exposed lower limbs below the knee, are disinfected with an iodophor cotton swab. Acupuncture points selected include GB34, GB39, BL60, BL40, ST41, KI9, and KI6. The practitioner applies pressure to the points with the left hand and swiftly inserts the needle with the right, using a 0.30mm*40mm disposable sterile acupuncture needle, penetrating the skin about 0.5-0.8 inches. After achieving deqi, the needle is twisted and thrust several times, left in place for 30 minutes. Upon removal, the needle site is compressed with a dry cotton swab until bleeding stops. Treatments occur every other day, totaling six sessions
  Interventions: Procedure: acupuncture

INTERVENTIONS:
Procedure: MNK therapy to release the superficial fascia — The patient, positioned supine and wearing shorts for full lower limb exposure, undergoes layered palpation by the practitioner at the procedure points, identifying tender nodules and swelling in superficial fascia and muscles, followed by disinfection with an iodophor cotton swab. The practitioner, donning sterile latex gloves, holds the micro-needle-knife between the thumb and index finger of the right hand, inserting it parallel to the body's longitudinal axis, while the left thumb presses and holds the cord-like nodules for parallel incisions, with a maximum insertion depth of 5mm, performing lifting and cutting motions. Depending on the nodule size, 1-3 incisions are made. Post-procedure, any bruising or tissue fluid is expelled by massaging from distal to proximal around the incision. The area is then compressed with dry sterile gauze until bleeding ceases. Treatments are administered every other day, totaling six sessions.
  Arms: Group 1 (MNK therapy to release the superficial fascia)
Procedure: acupuncture — Acupuncture treatment employing needles produced by Suzhou Medical Supplies Factory Co., Ltd., with specifications of 0.30mm*40mm and conforming to standard GB2024-1994. Patients, positioned prone or laterally with exposed lower limbs below the knee, are disinfected with an iodophor cotton swab. Acupuncture points selected include GB34, GB39, BL60, BL40, ST41, KI9, and KI6. The practitioner applies pressure to the points with the left hand and swiftly inserts the needle with the right, using a 0.30mm*40mm disposable sterile acupuncture needle, penetrating the skin about 0.5-0.8 inches. After achieving deqi, the needle is twisted and thrust several times, left in place for 30 minutes. Upon removal, the needle site is compressed with a dry cotton swab until bleeding stops. Treatments occur every other day, totaling six sessions
  Arms: Group 2 (acupuncture)

SUMMARY:
The goal of this type of randomized controlled trial, employing a blinded evaluator methodology, to verify the clinical efficacy and safety of MNK therapy. This aims to provide a reference for clinical practitioners and AAS patients in their decision-making process.

Participants will randomly allocated into two groups using a random number table method, with forty patients in each group. The experimental group (Group 1) underwent MNK therapy to release the superficial fascia, while the control group (Group 2) received conventional acupuncture treatment.

ELIGIBILITY:
Inclusion Criteria:

* 16 to 55 years old
* Clear history of trauma within 1 to 7 days
* Presence of localized swelling, pain, bruising, and limping symptoms in the ankle joint
* Pain in the ankle joint upon resistance
* No accompanying fractures
* Diagnosis of acute ankle injury according to the "Diagnostic and Therapeutic Criteria of Traditional Chinese Medicine"
* No prior treatment before participating in this therapy
* Willingness to participate in this study and signing of the informed consent form

Exclusion Criteria:

* Individuals with clear indications for surgery
* Those suffering from gout, rheumatoid arthritis, joint tuberculosis, joint tumors, etc.
* Pregnant or breastfeeding women
* Individuals with serious primary diseases of the cardiovascular, liver, kidney, brain, and hematopoietic systems
* Those with local skin lesions or skin diseases
* Individuals with coagulation dysfunction
* Those with severe fear of needles
* Individuals unwilling to comply with the treatment regimen

Ages: 16 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | up to one mont
  The VAS is utilized to assess the degree of pain experienced by the patient. Patients select an appropriate number (0 to 10) based on their perceived pain intensity: 0 indicates no pain and a normal state; 1 to 3 signifies mild pain that is tolerable and does not interfere with daily activities; 4 to 6 represents moderate pain that is noticeable and tolerable but affects daily life and sleep; 7 to 10 indicates severe pain that is intolerable.
Kofoed Ankle Score | up to one mont
  This score evaluates the functional recovery of the ankle joint following treatment, focusing on pain, function, and mobility. The total score is out of 100, with 85-100 classified as excellent, 75-85 as good, 70-74 as satisfactory, and below 70 as poor.

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-xiao Ma, Dr., Study Director — The Affiliated Dongyang Hospital of Wenzhou Medical University, Dongyang, Zhejiang, China
Locations (1):
- The Affiliated Dongyang Hospital of Wenzhou Medical University, Dongyang, Zhejiang, China, Dongyang, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No